CLINICAL TRIAL: NCT01165359
Title: A Randomized, Double-Blind, Phase 1b Study to Assess the Safety and Activity of the HCV Entry Inhibitor ITX 5061 in Treatment-Naive HCV Mono-Infected Adults
Brief Title: Evaluating the Safety of ITX 5061 in Treatment-Naive Hepatitis C (HCV)-Infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5277; 10836 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Part A: ITX 5061 (Experimental): Participants will receive ITX 5061 once a day for 3 days.
  Interventions: Drug: ITX 5061
- Part A: Placebo (Placebo Comparator): Participants will receive placebo once a day for 3 days.
  Interventions: Drug: Placebo ITX 5061
- Part B: ITX 5061 (Experimental): Participants will receive ITX 5061 once a day for 14 days.
  Interventions: Drug: ITX 5061
- Part B: Placebo (Placebo Comparator): Participants will receive placebo once a day for 14 days.
  Interventions: Drug: Placebo ITX 5061
- Part C: ITX 5061 (Experimental): Participants will receive ITX 5061 once a day for 28 days.
  Interventions: Drug: ITX 5061
- Part C: Placebo (Placebo Comparator): Participants will receive placebo once a day for 28 days.
  Interventions: Drug: Placebo ITX 5061

INTERVENTIONS:
Drug: ITX 5061 — For Part A of the study: 150 mg of ITX 5061, once a day for 3 days; 75 mg of ITX 5061, once a day for 3 days; or 25 mg of ITX 5061, once a day for 3 days.
  For Part B of the study: 150 mg of ITX 5061, once a day for 14 days; 75 mg of ITX 5061, once a day for 14 days; or 25 mg of ITX 5061, once a day for 14 days.
  For Part C of the study: 150 mg of ITX 5061, once a day for 28 days; 75 mg of ITX 5061, once a day for 28 days; or 25 mg of ITX 5061, once a day for 28 days.
  Arms: Part A: ITX 5061; Part B: ITX 5061; Part C: ITX 5061
Drug: Placebo ITX 5061 — For Part A of the study: placebo, once a day for 3 days.
  For Part B of the study: placebo, once a day for 14 days.
  For Part C of the study: placebo, once a day for 28 days.
  Arms: Part A: Placebo; Part B: Placebo; Part C: Placebo

SUMMARY:
Hepatitis C (HCV) is a disease that affects the liver. ITX 5061 is a new medication that is being tested to treat HCV. This study will evaluate the safety of ITX 5061 and examine different doses of the medication to evaluate which dose is the most effective at lowering the amount of HCV in the blood.

DETAILED DESCRIPTION:
HCV is a serious health concern and can lead to cirrhosis, liver cancer, and liver failure. Currently, HCV is treated with pegylated interferon and ribavirin, but these medications are not always effective and may have harmful side effects. ITX 5061 is a new medication that has been developed to treat HCV. This study will take place in three parts-Parts A, B, and C. Each part of the study will enroll participants for a different period of time, and within each part of the study, participants will receive varying amounts of ITX 5061. If ITX 5061 is found to be unsafe in any part of the study, the subsequent parts of the study will not occur. The purpose of this study is to evaluate the safety of different doses of ITX 5061 and determine the amount of time that is needed for ITX 5061 to safely lower the amount of HCV in the blood.

This study will enroll people with HCV who are HIV-uninfected. Participants will enroll in one of three parts of the study. They will be randomly assigned to receive ITX 5061 or placebo once a day for 3 days in Part A, for 14 days in Part B, or for 28 days in Part C. Within Parts A, B, and C, participants will receive either 150 mg, 75, mg, or 25 mg of ITX 5061. At a baseline study visit, participants will have a physical exam and blood and urine collection. All participants will receive their assigned medication at this visit. Participants in Part A will return for study visits on the 2 days after the baseline visit. During these study visits, participants will undergo a physical exam and will have blood collected several times over an 8-hour period. Participants in Part B of the study will attend study visits 1, 2, 3, 7, 10, and 13 days after the baseline visit. Participants in Part C of the study will attend study visits 1, 2, 3, 7, 10, 14, 21, and 27 days after the baseline visit. Participants in Parts B and C will undergo similar study procedures as participants in Part A. Throughout the study, participants will record their medication usage in a diary.

All participants will attend a study visit the day after they receive their last medication dose. In addition, participants in Part A will attend study visits 9 and 16 days after the baseline visit, participants in Part B will attend study visits 20 and 27 days after the baseline visit, and participants in Part C will attend study visits 34 and 41 days after the baseline visit. At each of these follow-up visits, participants will have a physical exam and a blood and urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Absence of HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit within 45 days prior to study entry
* Chronic HCV infection as defined and documented by testing. See protocol for details.
* HCV genotype 1 infection with source documentation from a College of American Pathologists (CAP) or Clinical Laboratory Improvement Amendments (CLIA) approved laboratory (or its equivalent) within 1 year prior to study entry. Those without a documented genotype result at screening will have a screening genotype performed either locally or provided by the study as described in the protocol.
* Serum or plasma HCV RNA greater than or equal to 100,000 IU/mL (5 log10) obtained within 45 days prior to study entry by any laboratory that has a CLIA certification or its equivalent
* Lack of significant hepatic fibrosis (bridging fibrosis or cirrhosis) confirmed by biopsy within 2 years of study entry or HCV FibroSURE score of less than or equal to METAVIR stage 2 within 1 year of study entry
* The following laboratory values obtained within 45 days prior to study entry:

  1. White blood cell (WBC) count greater than or equal to 3000/mm3
  2. Absolute neutrophil count (ANC) greater than or equal to 1000/mm3
  3. Hemoglobin greater than or equal to 12 g/dL for men and greater than or equal to 11 g/dL for women
  4. Platelet count greater than or equal to 120,000/mm3
  5. Alanine aminotransferase (ALT) less than or equal to 5 x the upper limit of normal (ULN)
  6. International normalized ratio (INR) less than 1.5
  7. Total bilirubin less than or equal to ULN
  8. Calculated creatinine clearance (CrCl) greater than or equal to 80 mL/min, as estimated by the Cockcroft-Gault equation. More information on this criterion can be found in the protocol.
* Hemoglobin A1c (HbA1c) less than or equal to 8.5% for participants with diabetes; must be obtained within 90 days prior to study entry
* Females of reproductive potential must have a negative serum or urine pregnancy test with a sensitivity of less than or equal to 25 mlU/mL within 45 days prior to study entry. More information on this criterion can be found in the protocol.
* All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization)
* If participating in sexual activity that could lead to pregnancy, participants must agree to use two reliable methods of contraception simultaneously while receiving study treatment and for 6 weeks after stopping study treatment. More information on this criterion can be found in the protocol.
* Participants who are not of reproductive potential are eligible to participate without requiring the use of contraceptives, with acceptable documentation of either sterilization or menopause required. More information on this criterion can be found in the protocol.
* Able and willing to provide written informed consent

Exclusion Criteria:

* Prior receipt of any interferon or ribavirin (RBV)
* Prior receipt of any therapy for HCV, including experimental treatments
* Evidence of decompensated liver disease manifested by presence of or history of ascites, variceal bleeding, or hepatic encephalopathy
* History of Gilbert's syndrome
* Presence of other known causes of significant liver disease including chronic or acute hepatitis B, acute hepatitis A, hemochromatosis, or homozygote alpha-1 antitrypsin deficiency
* History of known hepatocellular carcinoma
* History of major organ transplantation with an existing functional graft
* History of uncontrolled seizure disorders
* Breastfeeding
* Use of prohibited medications within 14 days prior to study entry. More information on this criterion can be found in the protocol.
* Initiation or change in dose of any nonprohibited prescription medication within 14 days prior to study entry
* Known allergy/sensitivity or any hypersensitivity to components of study drug or its formulation
* Any condition including active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 24 weeks prior to study entry; serious illness including malignancy, active coronary artery disease within 24 weeks prior to study entry; other chronic medical conditions that may preclude completion of the study in the clinical research site (CRS) investigator's opinion. Such conditions may be discussed with the protocol chair/vice chair (actgcorea5277@fstrf.org).
* Participation in a prior A5277 cohort

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Reduction in serum HCV RNA level greater than or equal to 1 log10 IU/mL from baseline at the end of treatment | Measured at the end of treatment (Day 3 in Part A, Day 14 in Part B, and Day 28 in Part C)
Adverse events (AEs) greater than or equal to grade 3 attributed to the study treatment by the cohort review group | Measured at the end of treatment (Day 3 in Part A, Day 14 in Part B, and Day 28 in Part C)

SECONDARY OUTCOMES:
Pharmacokinetic parameters (area under the curve [AUC], Cmax, Cmin) for ITX 5061 | Measured at the end of treatment (Day 3 in Part A, Day 14 in Part B, and Day 28 in Part C)
Quantitative change in HCV RNA from baseline at the study visits | Measured at the end of treatment (Day 3 in Part A, Day 14 in Part B, and Day 28 in Part C)
All reported AEs | Measured at the end of treatment (Day 3 in Part A, Day 14 in Part B, and Day 28 in Part C)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sulkowski, MD, Study Chair — Johns Hopkins University
Locations (10):
- United States (9):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico